CLINICAL TRIAL: NCT01180439
Title: Patient-Ventilator Interactions During Sleep Under Non-Invasive Ventilation in Severe Stable COPD
Brief Title: Patient-Ventilator Interactions in Chronic Obstructive Pulmonary Diseases (COPD) Under Non-Invasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Dan Adler, MD, Division of Pulmonary Diseases, Geneva University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CE 09-047
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Non-invasive ventilation; Chronic Obstructive Pulmonary Disease; Patient-ventilator synchronisation; Sleep study; Polysomnography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Adjustment of ventilator settings (device) — Decrease in pressure support, increase in respiratory back-up rate, increase in expiratory positive airway pressure (EPAP) to counteract effect of PEEPi, and adjustment of cycling (at higher percentage of peak inspiratory flow)

SUMMARY:
Non-invasive ventilation (NIV) in severe hypercapnic Chronic Obstructive Pulmonary Diseases (COPD) may be associated - during sleep - with recurrent episodes of patient ventilatory asynchrony, which in turn may affect quality of sleep, efficacy of ventilation and comfort of nocturnal NIV.Polysomnography (PSG) under NIV is necessary to detect these events.

Adjusting ventilator settings according to respiratory events detected by PSG with NIV may improve quality of sleep, efficacy of ventilation and comfort of nocturnal NIV.

DETAILED DESCRIPTION:
Patients under NIV for hypercapnic COPD have several reasons to develop patient-ventilatory asynchrony: delayed cycling, and insufficient expiratory time may induce progressive dynamic hyperinflation, and increase intrinsic positive end-expiratory pressure (PEEPi); too high levels of pressure support may also contribute to dynamic hyperinflation. Increase in PEEPi is associated with two respiratory events: unrewarded inspiratory efforts, and auto-triggering.

Our hypotheses are: 1/that these events occur frequently in COPD under NIV and that they are not detected by medical history or usual monitoring tools (SpO2; PtcCO2); 2/ that they can be easily detected by polysomnography; 3/ that simple adjustments of ventilator parameters aiming to reduce dynamic hyperinflation and unrewarded inspiratory efforts may improve efficacy of ventilation, quality of sleep and comfort of treatment.

The present study compares the results of two consecutive sleep studies: 1.PSG under NIV in severe stable COPD under "usual ventilator settings" with 2.PSG under NIV after adapting ventilator settings to results of initial PSG.

ELIGIBILITY:
Inclusion Criteria:

* COPD, with chronic hypercapnic respiratory failure, treated by NIV, in stable clinical condition, aged above 18 years

Exclusion Criteria:

* Unstable clinical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Subjective evaluation of efficacy of nocturnal ventilation after adjusting ventilator settings | one night
  Visual analogic scale (VAS) of morning dyspnea, and questionnaire evaluating 8 items of comfort of ventilation (Janssens JP et al; Impact of volume targeting on efficacy of bi-level non-invasive ventilation and sleep in obesity-hypoventilation; Respir Med 2009 Feb;103(2):165-72)

SECONDARY OUTCOMES:
Objective evaluation of efficacy of ventilation after adjustment of ventilator settings | one night
  Analysis of leaks, estimated ventilation, SpO2, TcPCO2, sleep structure, and patient-ventilatory synchronisation and comparison with data under "usual settings" for ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, MD, Study Director — Division of Pulmonary Diseases; Geneva University Hospital
Locations (1):
- Division of Pulmonary Diseases; Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Janssens JP, Metzger M, Sforza E. Impact of volume targeting on efficacy of bi-level non-invasive ventilation and sleep in obesity-hypoventilation. Respir Med. 2009 Feb;103(2):165-72. doi: 10.1016/j.rmed.2008.03.013. Epub 2008 Jun 24. PMID 18579368
- [Derived] Adler D, Perrig S, Takahashi H, Espa F, Rodenstein D, Pepin JL, Janssens JP. Polysomnography in stable COPD under non-invasive ventilation to reduce patient-ventilator asynchrony and morning breathlessness. Sleep Breath. 2012 Dec;16(4):1081-90. doi: 10.1007/s11325-011-0605-y. Epub 2011 Nov 4. PMID 22051930